CLINICAL TRIAL: NCT02111811
Title: Reducing the Burden of Depression on Employment: Improving Function and Work
Brief Title: Reducing the Burden of Depression Related Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1132-R; I01RX001132-01A1 (NIH)
Record Dates: First submitted 2014-03-31; First posted 2014-04-11 (Estimated); Results first posted 2020-04-08 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Depression
Keywords: Depression; Treatment Outcome; Delivery of Healthcare, Integrated; Employment; Rehabilitation
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Be Well At Work intervention + IC (Experimental): CBT based intervention focused on work productivity plus integrated care as usual
  Interventions: Other: Veterans Work and Health Initiative
- Integrated Care Only (No Intervention): usual care group (Behavioral Health lab care at the PVAMC)

INTERVENTIONS:
Other: Veterans Work and Health Initiative — CBT based intervention focused on work productivity
  Arms: Be Well At Work intervention + IC

SUMMARY:
The purpose of this research study is to test the effectiveness of a new telephone counseling program for employed Veterans with depression called the Veterans Work and Health Initiative (V-WHI) using the Be Well at Work (BWAW) intervention. 250 participants will be recruited and randomly assigned to one of two groups: the V-WHI experimental group or usual mental health care. The V-WHI counselors will address mental health and job-related issues that interfere with working. This counseling is provided solely over the phone with sessions every 2 weeks for 4 months (eight sessions total). At 8 months post-baseline, the V-WHI group is provided with a booster session. Participants in both groups are administered follow-up questionnaires at two time-points: month four and month nine.

DETAILED DESCRIPTION:
With the goal of helping employed Veterans with depression to participate fully in the labor market, this randomized controlled trial has two objectives: 1) test the effectiveness of a new evidence-based, vocationally-focused telephonic counseling program for employed Veterans with depression, the Veterans Work and Health Initiative (V-WHI), which was developed by this study's research partners from the Tufts Medical Center; and 2) if the V-WHI is effective, quantify its return on investment. This study will test the impact of the BWAW intervention in combination with the Philadelphia VA's Primary Care Mental Health Integration program, the Behavioral Health Lab (BHL).

For the main hypothesis, concerning the effect of BWAW, the primary endpoint is the post-intervention at-work mean productivity loss score based on the validated Work Limitation Questionnaire (WLQ) adjusted for baseline score. For Hypothesis 2, concerning maintenance of post-intervention effects at nine months, the primary outcome is the mean difference of the change in productivity loss score. For hypothesis 3, the primary outcome was the return on investment (ROI) from BWAW.

After informed consent and eligibility screening, subjects are randomized to one of two groups: the V-WHI intervention group or to the usual care group (BHL). 250 employed Veterans with depression and work limitations will be enrolled (half per group). The "usual care" group participants are assigned to standard behavioral health care. The second group, assigned to BWAW intervention, is the experimental group. Participants in this group are assigned to an innovative program designed explicitly to address mental health and vocational issues that interfere with working in addition to standard care. V-WHI counselors offer work coaching and modification strategies and work-focused cognitive behavioral therapy (CBT). This counseling is provided solely over the phone with sessions every 2 weeks for 4 months (eight sessions total). At 8 months post-baseline, the V-WHI group is provided with a booster session. Participants in both groups are administered follow-up questionnaires at two time-points: month four (post-intervention) and month nine.

ELIGIBILITY:
Inclusion Criteria:

Veterans will be considered eligible for study participation if the following criteria are met:

* 18 years of age (no maximum age is specified)
* working for pay 15 hours per week
* employed in the job for 6 months (to ensure that the Veteran has sufficient familiarity with the position and organization)
* current major depression and/or persistent depressive disorder symptoms based on DSM-5 criteria
* and current work limitations

Exclusion Criteria:

* Non-English speaking or reading
* bipolar disorder
* psychosis
* and/or planning to take maternity leave at any point in the next nine months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2014-05-19 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W. Oslin, MD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (2):
- United States (2):
  - Coatesville VA Medical Center, Coatesville, PA, Coatesville, Pennsylvania
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lerner D, Adler DA, Rogers WH, Ingram E, Oslin DW. Effect of Adding a Work-Focused Intervention to Integrated Care for Depression in the Veterans Health Administration: A Randomized Clinical Trial. JAMA Netw Open. 2020 Feb 5;3(2):e200075. doi: 10.1001/jamanetworkopen.2020.0075. PMID 32108889

RESULTS

PARTICIPANT FLOW:
Groups:
- Veterans Work and Health Initiative: Integrated care services plus a CBT based intervention focused on work productivity
  Veterans Work and Health Initiative: CBT based intervention focused on work productivity
- Integreated Care Only: usual care group (Integrated care services only)
Period: Treatment Phase
Arm/Group | Veterans Work and Health Initiative | Integreated Care Only
Started | 139 | 114
Completed | 115 | 96
Not Completed | 24 | 18
Not completed — Lost to Follow-up | 22 | 18
Not completed — Death | 2 | 0
Period: Follow up Period (Aim 2)
Arm/Group | Veterans Work and Health Initiative | Integreated Care Only
Started | 139 | 114 (All subjects were approached for followup, 1 patient completed the 2nd followup and not the first.)
Completed | 111 | 97
Not Completed | 28 | 17
Not completed — Lost to Follow-up | 26 | 17
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Veterans Work and Health Initiative | Integreated Care Only | Total
Number analyzed (Participants) | 139 | 114 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (11.6) | 44.8 (11.6) | 45.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 122 | 96 | 218
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 60 | 58 | 118
  White | 79 | 56 | 135
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 139 | 114 | 253
Depression Severity [Mean (Standard Deviation); unit: units on a scale] — PHQ9 is scored 0 to 27 with higher scores being greater distress. A change of 2 or more points is considered clinically relevant.
  units on a scale | 14.8 (4.8) | 14.1 (4.9) | 14.5 (4.8)
Work Productivity Lost Score [Mean (Standard Deviation); unit: units on a scale] — The WLQ scale ranges = 0 to 25. Higher scores indicate greater dysfunction. There are not specific cut off scores.
  units on a scale | 12.4 (4.9) | 12.3 (4.5) | 12.3 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Work Related Disability Post Intervention
Description: The outcome measure is the mean difference of the changes from baseline to time 1. The mean differences are then compared. The WLQ scale range=0-25 with higher scores indicating greater difficulty.
Time Frame: 4 months post randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Veterans Work and Health Initiative | Integreated Care Only
Number analyzed (Participants) | 115 | 96
units on a scale | -2.1 [-3.1 to -1.0] | -0.09 [-1.1 to 0.9]

2. Secondary Outcome: Sustained Improvement in Work Productivity
Description: The outcome measure is the mean difference of the changes from baseline until about 9 months post randomization. The mean differences are then compared. The WLQ scale range=0-25 with higher scores indicating greater difficulty.
Time Frame: 9 months post randomization
Population: There were more subjects available at 9 months than at the end of the trial (4 months) as we attempted to contact all patients who had not withdrawn. We were able to reach a few at 9 months who were not available at 4.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Veterans Work and Health Initiative | Integreated Care Only
Number analyzed (Participants) | 111 | 97
score on a scale | -3.4 [-4.5 to -2.3] | -.8 [-1.9 to 0.4]

3. Secondary Outcome: The Outcome is the Return on Investment (ROI) Obtained From Implementing the V-WHI Experimental Intervention.
Description: This variable is defined as: [marginal benefit on patient work productivity attributable to the V-WHI intervention] - [marginal cost of supplementing IC with V-WHI) / [marginal cost of supplementing IC with V-WHI]. The comparison assessed the monetized value of the difference in pre to post treatment changes in at-work productivity loss (presenteeism) + the monetized value of the difference in the changes in productivity loss due to work absences. Because both productivity loss components were measured at baseline and two follow-ups, the changes between time points (baseline to month 4 and month 4 to month 8/9) were first averaged before computing their difference.
  The marginal costs attributable to V-WHI included the full costs of the providing the counseling treatment and supervision of the counselors.
Time Frame: 9 months post randomization
Population: The marginal costs attributable to V-WHI included the full costs of the providing the counseling treatment and supervision of the counselors. The ROI analysis did not evaluate costs other than the V-WHI costs, including standard care provided to both the IC only group and the IC+V-WHI group.
Measure: Number; unit: marginal benefit in ($)
Arm/Group | Veterans Work and Health Initiative
Number analyzed (Participants) | 111
marginal benefit in ($) | 900

ADVERSE EVENTS:
Time Frame: 9 months of the trial
Description: Asked at the follow up assessments.
Arm/Group | Veterans Work and Health Initiative | Integreated Care Only
All-Cause Mortality (participants affected / at risk) | 2/139 | 0/114
Serious Adverse Events (participants affected / at risk) | 7/139 | 10/114
Other Adverse Events (participants affected / at risk) | 0/139 | 0/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Veterans Work and Health Initiative (N=139) | Integreated Care Only (N=114)
Hospitalization (Surgical and medical procedures) | 7 (7) | 10 (10) — Hospitalizations were identified through medical recorder review for dates of admission. We do not have information of the type hospitalization or the reason for hospitalization

LIMITATIONS AND CAVEATS:
This study includes data from one VHA medical center, which limits external validity. In addition, the sample size may have limited our power to detect some differences and we relied on self-report measures of occupational functioning.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT02111811/Prot_SAP_000.pdf